CLINICAL TRIAL: NCT04622579
Title: Lenalidomide Combined With Rituximab as Front-line Therapy in Elderly Patients Aged Over 80 Years With Diffuse Large B Cell Lymphoma
Brief Title: Lenalidomide Combined With Rituximab as Front-line Therapy for DLBCL Patients Aged Over 80 Years
Acronym: R2DLBCL80
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Guangzhou First People's Hospital (Other); First People's Hospital of Foshan (Other); Huizhou Municipal Central Hospital (Other); Shantou Central Hospital (Other)
Responsible Party: Principal Investigator, Wenyu Li, professor of medicine, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020099H
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B Cell Lymphoma; Age Over 80 Years
Keywords: lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lenalidomide combined with rituximab (Experimental): Rituximab 375 mg/m2 i.v d1 q28d； Lenalidomide 10mg Po. d1-21 q28d. After 6 cycles, patients obtained CR or PR will continue with Lenalidomide maintenance till the 24th month.
  Interventions: Drug: lenalidomide combined with rituximab

INTERVENTIONS:
Drug: lenalidomide combined with rituximab — lenalidomide and rituximab are dilivered as described, parameters concerning efficacy and safety are also obtained.

SUMMARY:
About 40% of Diffuse large B cell lymphoma relapse or is refractory, age is a prognostic factor of DLBCL, as elderly patients are not capable to received standard treatment, the prognosis of elderly patients is poor especially those aged over 80 years. In this study,we aimed to investigate the safety and efficacy of the combination of lenalidomide and rituximab in elderly patients aged ≥ 80 years with untreated DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧80 years ;
2. ECOG score 0-2；
3. untreated with pathologically conﬁrmed CD20+ DLBCL ;
4. expected life expectancy of ≥ 12 weeks;
5. capable of swallowing tablets;
6. GFR(by Cockcroft- Gault)≥30 ml/min;
7. can sign written informed consent to participate in the study.

Exclusion Criteria:

1. with CNS involvement;
2. with other malignancy (not including adequate-treated non-melanoma cutaneum carcinoma); patients with other cancer but disease-free for ≥5 years can enter this study;
3. with ≥ grade 2 peripheral neurophathy;
4. with cardiopathy including unstable angia or myocardial infarction over the past 8 weeks;
5. received live vaccine within 28 days.;
6. HIV-positive;
7. thrombosis ;
8. GFR<30 mL/min;
9. other conditions not suitable for rituximab or lenalidomide application.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  Overall response rate

SECONDARY OUTCOMES:
CR | 24 months
  Complete response
OS | from date of treatment until the date of death from any cause, assessed up to 5 years
  Overall survival
PFS | from date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China